CLINICAL TRIAL: NCT05209230
Title: Is Myocardial Stunning Induced by Continuous Renal Replacement Therapy a Reality in Critically Ill Patients?
Acronym: MS-CRRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69HCL21_1013
Record Dates: First submitted 2022-01-11; First posted 2022-01-26 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Acute Kidney Injury KDIGO 3; Continuous Renal Replacement Therapy Initiated by the Clinician in Charge Without Emergency; Myocardial Stunning
Keywords: Acute kidney injury,; continuous renal replacement therapy; myocardial stunning; regional wall motion abnormalities; 2D speckle tracking echocardiography
MeSH Terms: conditions — Myocardial Stunning; Acute Kidney Injury | interventions — Continuous Renal Replacement Therapy; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous renal replacement therapy arm (Experimental): Echocardiographic evaluation (with 2D speckle tracking analysis of left ventricular segmental function) 1 hour before and 3 hours after the initiation of continuous renal replacement therapy (continuous veno venous hemofiltration) initiation
  Interventions: Procedure: Continuous renal replacement therapy
- Control arm (Other): Two echocardiographic evaluations (with 2D speckle tracking analysis of left ventricular segmental function) at an interval of 4 hours, before the continuous renal replacement therapy initiation.
  Interventions: Other: Control group

INTERVENTIONS:
Procedure: Continuous renal replacement therapy — Continuous renal replacement therapy (veno venous hemofiltration) without net ultrafiltration, through a dedicated central venous catheter
  Arms: Continuous renal replacement therapy arm
Other: Control group — Continuous renal replacement therapy is differed from 6 hours to allowed 2 control echocardiographic evaluations
  Arms: Control arm

SUMMARY:
Myocardial stunning during chronic intermittent hemodialysis is a well-described phenomenon. Little case series of patients presenting myocardial stunning during renal replacement therapy for acute kidney injury in critically ill patients are reported, with intermittent hemodialysis and continuous renal replacement therapy. However, the small sample sizes and the absence of a control arm limit their interpretation, mainly whether the myocardial stunning may be related to cardiac loading conditions variations and whether it may impact the hemodynamic.

The investigator hypothesize that myocardial stunning induced by renal replacement therapy is frequent, independent from cardiac loading conditions and associated with peripheral hypoperfusion.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Acute Kidney Injury grade 3 (KDIGO)
* Indication for renal replacement therapy for the clinician in charge

Exclusion Criteria:

* Emergency indication to renal replacement therapy (pH<7.15, Kaliemia > 6mmol/L, refractory pulmonary oedema)
* Poor echogenicity with speckle tracking analysis failure
* Chronic hemodialysis
* Extra corporeal membrane oxygenation, left ventricular assist device.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2025-12-18 (Actual); Study Completion 2025-12-18 (Actual)

PRIMARY OUTCOMES:
Number of segment of the left ventricle with regional wall motion abnormalities | Change between the echocardiography at baseline and the echocardiography 4 hours after.
  Numbers of segments of the left ventricle (by patient) with a decrease greater than 20% of the peak systolic longitudinal strain (2D speckle tracking) on the second echocardiography as compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: RUSTE Martin, MD, Msc, Principal Investigator — Hospices Civils de Lyon
Locations (3):
- France (3):
  - Département d'anesthésie-réanimation Hôpital cardiologique Louis Pradel Groupe Hospitalier Est, Bron, Bron
  - Ruste Martin, Bron, BRON
  - Hopital Edourd Herriot, Lyon